CLINICAL TRIAL: NCT04474834
Title: GENetic Risk Estimation of Breast Cancer Prior to Decisions on Preventive Therapy Uptake, Risk Reducing Surgery or Intensive Imaging Surveillance: A Study to Determine if a Polygenic Risk Score Influences the Decision Making Options Amongst High Risk Women (GENRE 2)
Brief Title: Genetic Risk Estimations for Influencing Decision Making in Women at High Risk of Breast Cancer, GENRE 2 Study
Acronym: GENRE2
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sandhya Pruthi, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 19-003085; NCI-2022-02838 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: BCRAT; IBIS; Breast Cancer; BRCA1; BRCA2; BRCA; BRCA 1/2; Tyrer-Cuzick; CEDM; PRS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants indicate yes/no on consent form regarding retention of blood samples with DNA for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PRS: Providing polygenic risk score (PRS)
  Interventions: Genetic: Polygenic Risk Score

INTERVENTIONS:
Genetic: Polygenic Risk Score — A Polygenic Risk Score (PRS) is a blood based genetic test which assesses 300 common breast cancer susceptibility loci (Single Nucleotide Polymorphisms). The PRS has been retrospectively validated and categorizes women into three categories of lifetime risk of developing breast cancer: Low Risk (<15% lifetime risk), Above Average Risk (15 to 40%), and high risk (>40 %).

SUMMARY:
The primary aim of this study is to determine if the addition of an individual polygenic risk score (PRS) in addition to the Breast Cancer Risk Assessment Tool (BCRAT) or Tyrer-Cuzick (IBIS) score will aid women at risk of breast cancer in making a decision to take (or not take) medications to prevent breast cancer.

DETAILED DESCRIPTION:
This is a minimal risk prospective multisite study with a single arm incorporating the PRS into a standard breast cancer risk reduction consultation, followed by annual surveys over 10 years to determine if and how the availability of the PRS influenced patient decisions regarding preventive medicine and medication compliance. Because women know beforehand that the PRS is pending, study participants will be advised that a final decision to take preventive medicine must be deferred until after the PRS results are made available. Nevertheless, a survey of understanding of risk and benefit and assessment of willingness to take preventive medicine will be done prior to receiving the PRS results and then another survey will be completed after receiving the PRS score.

ELIGIBILITY:
Inclusion Criteria:

* Women >= 35 years old and =< 75 years old with at least one of the following:

  * A National Cancer Institute (NCI)-BCRAT 5 year risk of >= 3% which corresponds to the level in which there is moderate evidence of treatment benefit outweighing risk according to the United States (US) Preventative Services Task Force
  * IBIS (Tyrer-Cuzik) score for the 10 year risk of breast cancer of >= 5%
  * History atypical ductal hyperplasia or atypical lobular hyperplasia with a BCRAT >= 3% or IBIS >= 5%
  * History of lobular carcinoma in situ with a BCRAT >= 3% or IBIS >= 5% OR
* Women >= 18 years old or =< 75 years old with a BRCA 1 or 2 mutation, CHEK 2, PALB 2, ATM, or other hereditary breast mutation carrier per investigator
* Willing and able to provide an email address to receive study surveys
* Able to participate in all aspects of the study
* Understand and sign the study informed consent

Exclusion Criteria:

* Women whose BCRAT falls below the threshold (<3 % 5 year risk) of moderate benefit according to the US Preventative Task Force AND Women whose IBIS score is <8% for the 10 year risk
* Women with known contra-indications to Tamoxifen, raloxifene ,exemestane, or anastrazole
* Current or prior use of Tamoxifen, raloxifene, exemestane or anastrazole
* Unable to give informed consent
* Prior history of invasive breast cancer, ductal carcinoma in situ or other breast cancers
* At high risk due to prior radiation therapy to the chest
* Women who are pregnant or breastfeeding
* Prior risk reducing or prophylactic mastectomy
* Unwilling or unable to provide an email address for study surveys to be sent to
* Subject has a known history or any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women attending the Mayo Clinic Breast Cancer clinics in Rochester, Arizona and Florida or the Mayo Clinic Health System in Austin or Albert Lea who meet eligibility criteria will be offered participation in this study after initial clinical calculation of the BCRAT or IBIS score and counseling as to the advisability of preventive therapy.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient self-reported intention to take a breast cancer preventing medication | up to 6 months after initial consultation

SECONDARY OUTCOMES:
Proportion of patients who are taking preventative medications each year for 10 years | Each year for up to 10 years
Endocrine related quality of life scores each year for 10 years | Each year for up to 10 years
Proportion of patient who are pursuing supplemental screening for 10 years | Each year for up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Pruthi, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University, Evanston, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials